CLINICAL TRIAL: NCT06023459
Title: Randomized Controlled Pilot Trial of Extended-released Buprenorphine vs. Sublingual Buprenorphine-naloxone in Rural Settings
Brief Title: Extended-release Buprenorphine Compared to Sublingual Buprenorphine in Rural Settings (RXR)
Acronym: RXR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yih-Ing Hser (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH); The Emmes Company, LLC (Industry); University of California, Los Angeles (Other); RAND (Other); Cornell University (Other); Oregon Health and Science University (Other); University of Illinois at Chicago (Other); University of Washington (Other); West Virginia University (Other)
Responsible Party: Sponsor-Investigator, Yih-Ing Hser, Distinguished Research Professor, Department of Psychiatry and Behavioral Sciences, Geffen School of Medicine, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN-0102-XR; UG1DA049435 (NIH)
Record Dates: First submitted 2023-08-08; First posted 2023-09-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders; Narcotic-Related Disorders
Keywords: Opioid Use Disorder; Opioid Medication Assisted Treatment; Buprenorphine; Comparative Effectiveness Research
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Narcotic-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: A 24-month randomized controlled open-label pilot study will be conducted in approximately 6 clinics in rural settings. Participants will be randomized within each clinic to XR-BUP or SL-BUP in a ratio of 2:1 (overall approximately 96 in the XR-BUP condition, 48 in the SL-BUP condition). They will receive study medication for approximately 14 weeks following randomization, including an initial ~2-week period of induction/stabilization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Injectable extended-release buprenorphine (XR-BUP) (Experimental): Participants will be randomly assigned to XR-BUP, with approximately 96 in the XR-BUP condition. The XR-BUP condition will use Brixadi/CAM2038 injectable, extended-release buprenorphine (Braeburn Pharmaceuticals, Inc.). After titrating to a stable dosage in approximately two weeks using weekly injection dosages as clinically indicated to relieve cravings and withdrawal symptoms, the target monthly dosage (128mg) of XR-BUP will be administered by injection at approximately Day 14 and approximately four weeks later in Week 6, with a third injection in Week 10. Dosage adjustments will be made as indicated for tolerability.
  Interventions: Drug: Injectable extended-release buprenorphine
- Sublingual buprenorphine-naloxone (SL-BUP) (Active Comparator): Participants will be randomly assigned to SL-BUP with approximately 48 in the SL-BUP condition. The SL-BUP condition will use sublingual buprenorphine-naloxone, with a target maintenance daily dose range of 16-24mg as recommended for clinical practice. Titration to maintenance dosage will be attempted within the first two weeks of the SL-BUP condition. During the initial stabilization weeks, SL-BUP will be flexibly dosed as clinically indicated to relieve cravings and withdrawal symptoms, after which dosage adjustments will be based on clinical decisions by the site clinicians. The maintenance dosage of SL-BUP will be dispensed on a schedule similar to the XR-BUP injections (i.e., at approximately Day 14, Week 6, and Week 10).
  Interventions: Drug: Sublingual buprenorphine-naloxone

INTERVENTIONS:
Drug: Injectable extended-release buprenorphine — Participants randomized to the XR-BUP condition will receive XR-BUP study medication for approximately 14 weeks following randomization, including an initial ~2-week period of induction/stabilization.
  Other Names: XR-BUP (Brixadi)
  Arms: Injectable extended-release buprenorphine (XR-BUP)
Drug: Sublingual buprenorphine-naloxone — Participants randomized to the SL-BUP condition will receive SL-BUP study medication for approximately 14 weeks following randomization, including an initial ~2-week period of induction/stabilization.
  Other Names: SL-BUP
  Arms: Sublingual buprenorphine-naloxone (SL-BUP)

SUMMARY:
This pilot trial will explore the feasibility, acceptability, and effectiveness of the most recently approved formulation of injectable extended-release buprenorphine (XR-BUP) for treatment of opioid use disorder (OUD) in rural settings. We will randomize 144 eligible individuals with moderate to severe OUD in a 2:1 ratio to one of two medication conditions: (1) XR-BUP (128mg target), administered every 4 weeks or (2) SL-BUP (16mg-24 mg/day target).Participants will receive study medication treatment for the 14 week-intervention period, including an initial ~2-week period of induction/stabilization. The study will use a mixed-methods approach (participant assessments, study medication records, qualitative interviews) for assessing feasibility and acceptability, and results will include patient outcome data on the comparative effectiveness of XR-BUP versus SL-BUP for patients with OUD in rural settings.

DETAILED DESCRIPTION:
This 24-month randomized controlled open-label pilot study will be conducted in approximately 6 clinics in rural settings. The study objectives are to describe the feasibility of implementing the study in rural settings, document the acceptability of the XR-BUP condition, and assess the comparative effectiveness of XR-BUP compared with SL-BUP. Participants will be randomized within each clinic to XR-BUP or SL-BUP in a ratio of 2:1 (overall approximately 96 in the XR-BUP condition, 48 in the SL-BUP condition). They will receive study medication for approximately 14 weeks following randomization, including an initial ~2-week period of induction/stabilization. The XR-BUP condition will use Brixadi®/CAM2038 injectable, extended-release buprenorphine. The measure for the main comparative effectiveness outcome is number of urine drug screen (UDS) results negative for opioids at scheduled assessments during Week 2 through Week 14 of the trial. Missing or positive UDS for any non-prescribed opioid is considered UDS positive.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age
2. Meet DSM-5 criteria for moderate to severe OUD or be on buprenorphine medication for OUD
3. Be interested in receiving buprenorphine treatment for OUD
4. Be willing to be randomized to either SL-BUP or XR-BUP
5. Be willing to comply with all study procedures
6. Be in good general health, as determined by the study Medical Clinician based on medical/psychiatric histories and physical exam, to permit treatment in an outpatient setting
7. If female of childbearing potential, be willing to practice an effective method of birth control for the duration of participation in the study intervention and agree to study-administered pregnancy testing during their participation in the study
8. Be able to speak English sufficiently to understand the study procedures
9. Be willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

1. Have evidence of a serious psychiatric disorder as assessed by the study Medical Clinician that would make participation difficult or unsafe (e.g., active psychosis, severe depression, or mania)
2. Have suicidal or homicidal ideation or behavior that requires immediate attention
3. Have a medical condition or serious medical illness that, in the opinion of the study Medical Clinician, would make study participation medically unsafe
4. Have been in treatment with naltrexone within 28 days of consent
5. Have been in methadone maintenance treatment within 28 days of consent
6. Be taking medication or require any medication that, in the judgment of the study Medical Clinician, could interact adversely with study medication
7. Have known allergy or sensitivity to SL-BUP or XR-BUP formulations or their components
8. Be currently incarcerated or have pending legal action that could preclude participation in study activities
9. Have other situation that might prevent the participant from remaining in the area for the duration of the study (e.g., planned move)
10. Have a current pattern of alcohol, benzodiazepine, or other sedative hypnotic use, as determined by the study Medical Clinician, that would require a different level of care and preclude safe participation in the study
11. Be currently pregnant or breastfeeding or planning on conception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Comparative effectiveness | Week 2 through Week 14 of the trial
  Number of urine drug screen (UDS) results negative for opioids
Feasibility of study implementation | 14 weeks of the trial starting at randomization
  The extent to which XR-BUP can be implemented in rural clinic settings, including recruitment, consent, study completion.
Acceptability | 14 weeks of the trial starting at screening
  Acceptability of XR-BUP by those implementing or receiving XR-BUP if it is agreeable or satisfaction, percent receiving the first monthly injection, percent receiving at least the first two monthly injection

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Ing Hser, PhD, Principal Investigator — University of California, Los Angeles; Larissa Mooney, MD, Principal Investigator — University of California, Los Angeles
Locations (7):
- United States (7):
  - AppleGate Recovery El Dorado, El Dorado, Arkansas
  - Southern Humboldt Community Healthcare District - Jerold Phelps Community Hospital, Garberville, California
  - Gibson Area Hospital and Health Services - Gibson Recovery Optimizing Wellness, Gibson City, Illinois
  - Penobscot Community Health Care Inc. - Seaport Community Health Center, Belfast, Maine
  - Oregon Health & Science University Primary Care Clinic, Scappoose, Scappoose, Oregon
  - Providence Northeast Washington Medical Group, Colville, Washington
  - New Beginnings Recovery Clinic & Behavioral Health Center, New Martinsville, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Implementation Guidance and the HEAL Public Access and Data Sharing Policy. Primary data for this study will be available to the public in the NIDA Data Share repository, per NIDA CTN policy. For more details on data sharing please visit https://datashare.nida.nih.gov/.The main outcome(s) publication will be included along with study underlying primary data in the data share repository, and it will also be deposited in PubMed Central http://www.pubmedcentral.nih.gov/ per NIH Policy (http://publicaccess.nih.gov/).
Time Frame: After the main outcome(s) paper(s) have been published or 18 months after data lock, whichever comes first.
Access Criteria: For more details on data sharing please visit https://datashare.nida.nih.gov
URL: https://datashare.nida.nih.gov